CLINICAL TRIAL: NCT02445508
Title: Effect of Bile Acid Secretion and Sequestration on GLP-1 Secretion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Andreas Brønden, MD, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NCT02445508
Record Dates: First submitted 2015-05-08; First posted 2015-05-15 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sevelamer; Cholecystokinin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo+Placebo (Placebo Comparator): Oral ingestion of sevelamer placebo powder combined with intravenous infusion of isotonic saline.
  Interventions: Drug: Sevelamer placebo; Drug: Isotonic saline
- Placebo+Cholecystokinin (Active Comparator): Oral ingestion of sevelamer placebo powder combined with intravenous infusion of cholecystokinin.
  Interventions: Drug: Cholecystokinin; Drug: Sevelamer placebo
- Sevelamer+Placebo (Active Comparator): Oral ingestion of sevelamer powder combined with intravenous infusion of isotonic saline.
  Interventions: Drug: Sevelamer; Drug: Isotonic saline
- Sevelamer+Cholecystokinin (Active Comparator): Oral ingestion of sevelamer powder combined with intravenous infusion of cholecystokinin.
  Interventions: Drug: Sevelamer; Drug: Cholecystokinin

INTERVENTIONS:
Drug: Sevelamer
  Arms: Sevelamer+Cholecystokinin; Sevelamer+Placebo
Drug: Cholecystokinin
  Arms: Placebo+Cholecystokinin; Sevelamer+Cholecystokinin
Drug: Sevelamer placebo
  Arms: Placebo+Cholecystokinin; Placebo+Placebo
Drug: Isotonic saline
  Arms: Placebo+Placebo; Sevelamer+Placebo

SUMMARY:
Accumulating evidence suggests that bile acids in our intestines may constitute essential components in the complex mechanisms regulating gut hormone secretion and glucose homeostasis. Thus, it is likely that modification of the enterohepatic circulation of bile acids can lead to changes in gut hormone secretion and consequently affect glucose homeostasis.

The current study is a human interventional randomized controlled cross-over study including four study days for each participant. As a tool to sequester bile acids we will use sevelamer, a phosphate binding resin used in the treatment of hyperphosphataemia in adult patients with chronic kidney disease. Surprisingly, sevelamer has been shown to improve glycaemic control in patients with chronic kidney disease and type 2 diabetes. Intravenous infusion of cholecystokinin will be used to elicit gallbladder contraction and emptying. The aim is to examine how (and if) bile acid sequestration can influence postprandial glucagon-like peptide-1 (GLP-1) secretion and glucose homeostasis in patients with type 2 diabetes.

The investigators hypothesize that higher luminal concentrations of bile acids in the distal gut will elicit changes in gut hormone secretion. The current study will help to clarify this hypothesis and improve our general understanding of the association between bile acid circulation and signalling, gut hormone secretion and glucose metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least 3 months (diagnosed according to the criteria of the World Health Organization (WHO))
* Men and postmenopausal women
* Metformin applied as the only anti-diabetic drug
* Caucasian ethnicity
* Normal haemoglobin
* Age above 40 years and below 70 years
* BMI >23 kg/m2 and <35 kg/m2
* Informed and written consent

Exclusion Criteria:

* Liver disease (alanine aminotransferase (ALAT) and/or serum aspartate aminotransferase (ASAT) >2 times normal values) or history of hepatobiliary disorder
* Gastrointestinal disease, previous intestinal resection, cholecystectomy or any major intra-abdominal surgery
* Nephropathy (serum creatinine >150 µM and/or albuminuria)
* Hypo- and hyperthyroidism
* Hypo- and hypercalcaemia
* Hypo- and hyperphosphataemia
* Active or recent malignant disease
* Treatment with medicine that cannot be paused for 12 hours
* Treatment with oral anticoagulants
* Any treatment or condition requiring acute or sub-acute medical or surgical intervention
* Any condition considered incompatible with participation by the investigators

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Glucagon-like peptide-1 (GLP-1): Incremental and total area under the Concentration-Time Curve | -30, -15, 0, 10, 20, 30, 45, 60, 90, 120, 180, 240 min on study days 1-4
  Incremental and total area under the Concentration-Time Curve (AUC 0-240 min)

SECONDARY OUTCOMES:
Responses of various other gut hormones: Incremental and total area under the Concentration-Time Curve | -30, -15, 0, 10, 20, 30, 45, 60, 90, 120, 180, 240 min on study days 1-4
  Incremental and total area under the Concentration-Time Curve (AUC 0-240 min)
Blood analysis of paracetamol as an assessment of gastric emptying | -30, -15, 0, 10, 20, 30, 45, 60, 90, 120, 180, 240 min on study days 1-4
  Assessment of gastric emptying
Indirect calorimetry: Basal metabolic rate | -30 min to 240 min
  Basal metabolic rate
Gallbladder volume as assessed by Ultrasound measurements | -30 min to 240 min
  Gallbladder volume
Appetite as assessed by Visual analog scale score | -30 min to 240 min
  Appetite

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Diabetes Research, Hellerup, Denmark